CLINICAL TRIAL: NCT05863039
Title: Resistance Training With Blood Flow Restriction for the Lower Extremity Muscles
Brief Title: Resistance Training With Blood Flow Restriction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14083
Record Dates: First submitted 2023-04-17; First posted 2023-05-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: resistance training; strength training; blood flow restriction; motor units; body composition
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Strength training associated with blood flow restriction
  Interventions: Other: Blood flow restriction
- Group 2 (Experimental): Conventional strength training using high loads
  Interventions: Other: Regular training type 1
- Group 3 (Experimental): Conventional strength training using low loads
  Interventions: Other: Regular training type 2

INTERVENTIONS:
Other: Blood flow restriction — Strength training of the lower leg muscles using blood flow restriction
  Arms: Group 1
Other: Regular training type 1 — Strength training of the lower leg muscles using high loads
  Arms: Group 2
Other: Regular training type 2 — Strength training of the lower leg muscles using low loads
  Arms: Group 3

SUMMARY:
Blood flow restriction associated with resistance training is suggested to potentiate increases in muscular strength and hypertrophy. This study will compare the effects of resistance training associated with blood flow restriction with a regular resistance training program. Findings of this project will provide important information regarding a promising intervention to potentiate muscle performance.

DETAILED DESCRIPTION:
The purpose of this study is to determine alterations in motor unit behavior of the tibialis anterior muscles after a resistance exercise program associated with blood flow restriction. Our working hypothesis is that blood flow restriction to working muscles will induce greater changes in muscle activation, lean mass and muscle size compared with a training at same intensity without blood flow restriction.

ELIGIBILITY:
Exclusion Criteria:

* presence of neurological diseases,
* presence of metal implants or joint replacement
* any restriction to perform physical activity
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Force | 10 sessions (up to 6 weeks)
  Force of the lower leg muscles using a custom made ergometer

SECONDARY OUTCOMES:
Body composition | Start and end of the protocol
  dual x-ray absorptiometry (DEXA) will be used to assess body composition

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Pereira, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified information can be shared according to instructions of the local institutional review board that reviewed the study
Supporting Information: Study Protocol